CLINICAL TRIAL: NCT07339540
Title: Clinical Study on the Safety and Efficacy of Targeted BCMA In Vivo LV Injection in the Treatment of Recurrent or Refractory Autoimmune Diseases
Brief Title: the Safety and Efficacy of Targeted BCMA In Vivo LV Injection for Recurrent or Refractory Autoimmune Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Lingli Dong, professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRG2503E2
Record Dates: First submitted 2025-11-26; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Recurrent or Refractory Systemic Lupus Erythematosus; Recurrent or Refractory IgG4 Related Diseases; Recurrent or Refractory Systemic Sclerosis; Recurrent or Refractory Idiopathic Inflammatory Myopathy; Recurrent or Refractory ANCA Associated Vasculitis
MeSH Terms: conditions — Recurrence; Lupus Erythematosus, Systemic; Immunoglobulin G4-Related Disease; Scleroderma, Systemic; Myositis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V001-BCMA injection (Experimental)
  Interventions: Drug: V001-BCMA

INTERVENTIONS:
Drug: V001-BCMA — Targeted BCMA In-vivo LV Injection (Code: V001-BCMA) is a third-generation non-replicating self-inactivating lentiviral vector. Its envelope protein has been engineered to express targeting molecules on the lentiviral surface for specific recognition of T cells, while its nucleic acid contains a T cell-specific promoter and a CAR gene. After specifically targeting and binding to T cells, V001-BCMA enables the expression of CAR on the surface of T cells, forming CAR-T cells. These CAR-T cells can then specifically kill target cells.

SUMMARY:
This study is designed as a single arm, open label, single center clinical trial to evaluate the safety, tolerability, efficacy, pharmacokinetic or pharmacodynamic characteristics of the investigational drug V001-BCMA in autoimmune disease.

ELIGIBILITY:
Inclusion Criteria:

* 1. The age at the time of signing the informed consent form is ≥18 years old and ≤65 years old;
* 2. For cohort 1: recurrent or refractory systemic lupus erythematosus (all of the following four items must be met simultaneously)

  1. Diagnosed with SLE according to the 2012 SLICC or 2019 EULAR/ACR revised criteria.
  2. During screening, the patient exhibits positive anti-nuclear antibodies, and/or positive anti-ds-DNA antibodies, and/or positive anti-Smith antibodies.
  3. Before screening, patients must have received treatment with glucocorticoids combined with immunosuppressants and/or biologics for at least 3 months, with a stable dose for more than 2 weeks, and the disease remains active or the patient is intolerant to the medication.
  4. During the screening period, the SLEDAI-2K score is ≥8 points
* 3. For cohort 2: recurrent or refractory IgG4-related disease (all three of the following criteria must be met simultaneously)

  1. Meet the American College of Rheumatology (ACR)/EULAR 2019 classification criteria for IgG4-RD.
  2. Patients with clinical manifestations of recurrent or refractory IgG4-RD and ineffective conventional treatment
  3. Meet the clinical phenotype of "Mikulicz-system involvement"
* 4. For cohort 3: relapsed or refractory systemic sclerosis (all of the following 5 items must be met simultaneously)

  1. Meet the 2013 American College of Rheumatology (ACR) and European League Against Rheumatism (EULAR) classification criteria for SSc.
  2. Anti-Scl 70 antibody positive, or anti-centromere protein antibody positive, or anti-RNA polymerase III antibody positive
  3. Patients with a modified Rodnan skin score (mRSS) of ≥10 at screening
  4. Before screening, patients must have received treatment with glucocorticoids combined with immunosuppressants and/or biologics for at least 3 months, with a stable dose for more than 2 weeks, and the disease remains active or intolerable.
* 5. For cohort 4: relapsed or refractory idiopathic inflammatory myopathies (all of the following 5 criteria must be met)

  1. Meet the 2017 EULAR/ACR classification criteria for inflammatory myopathies (including dermatomyositis DM, polymyositis PM, anti-synthetase syndrome ASS, and necrotizing myositis NM).
  2. At least one myositis-specific antibody (MSA) or myositis-associated antibody (MAA) positive (+ or above)
  3. During the screening period, the patient meets 2 of the following criteria: PGA(VAS)≥2cm (VAS-10cm scale); PtGA(VAS)≥2cm (VAS-10cm scale); HAQ>0.25; one or more muscle enzymes are elevated (CK, LDH, AST, ALT) ≥1.5×ULN; overall muscle extrinsic assessment (MDAAT) ≥2.0cm (VAS-10cm scale)
  4. After at least 3 months of treatment with glucocorticoids and immunosuppressants and/or biologics, with stable doses for more than 2 weeks, the disease remains active or the patient is intolerant to the medication.
  5. Active myositis is present in muscle biopsy or muscle MRI during the screening period or within the first 6 months before the screening period.
* 6. For cohort 5: relapsed or refractory AAV (all three of the following conditions must be met simultaneously)

  1. According to the 2022 ACR/EULAR criteria, the patient is diagnosed with AAV (GPA or MPA subtype). According to the KDIGO guidelines, after 3 months of treatment with glucocorticoids combined with immunosuppressants such as cyclophosphamide or biologics such as rituximab, and the dose is stable for more than 2 weeks, the disease is still active or the patient is intolerant to the drug;
  2. The patient is currently or has been in the course of AAV related antibodies positive;
  3. Severe disease requiring treatment (BVAS score ≥3.0).
* 7. Possess sufficient organ function
* 8. Men with fertility and women of childbearing age must agree to use effective contraception from the time they sign the informed consent form until 1 year after the study drug is administered. Blood pregnancy tests for women of childbearing age must be negative at screening and before infusion;
* 9. The subject or his/her guardian agrees to participate in this clinical study and signs the informed consent form (ICF), indicating that he/she understands the purpose and procedures of this clinical study and is willing to participate in the study.

Exclusion Criteria:

* 1. For cohort 1: relapsed or refractory systemic lupus erythematosus

  1. Subjects with uncontrolled lupus crisis within 8 weeks before screening were assessed by the investigator as unsuitable for participation in this study.
  2. Before screening, patients with clinically significant central nervous system diseases or pathological changes not caused by lupus, including but not limited to cerebrovascular accident, aneurysm, epilepsy, convulsion/convulsion, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, brain organic syndrome, or mental illness, should be excluded.
* 2. For cohort 3: relapsed or refractory systemic sclerosis. High-risk pulmonary arterial hypertension, according to the "Risk Stratification of Arterial Pulmonary Arterial Hypertension (PAH)" in the "Guidelines for the Diagnosis and Treatment of Pulmonary Arterial Hypertension in China (2021 Edition)".
* 3. History of major organ transplantation (such as heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation.
* 4. Subjects with a history of ≥ Grade 2 bleeding within 30 days prior to screening, as assessed by the investigator, were deemed unsuitable for enrollment.
* 5. Use of any live vaccines against infectious diseases within 8 weeks before infusion.
* 6. Received any treatment using vesicular stomatitis virus G (VSVG) pseudotype virus.
* 7. The subject has a history or evidence of suicidal thoughts within 6 months before signing the ICF, or any suicidal behavior within 12 months before signing the ICF, and the researcher believes that there is a significant risk of suicide.
* 8. Pregnant or lactating women;
* 9. The patient has a history of severe and/or uncontrolled liver, gastrointestinal, kidney, lung, cardiovascular, psychiatric, neurological, or musculoskeletal diseases, hypertension, or any other medical condition that, in the opinion of the investigator, may affect the integrity of the patient's participation in the study, or may endanger the safety of the subject or affect the validity of the study results.
* 10. Suffered from malignant tumor within 3 years before screening, except for the following conditions: received radical treatment for malignant tumor and had no known active disease within ≥3 years before enrollment; or had fully treated non-melanoma skin cancer and currently had no evidence of disease;
* 11. Received any B-cell depleting biologic therapy (e.g., rituximab, ocrelizumab, obinutuzumab, ofatumumab, inebilizumab, etc.) within 3 months prior to infusion, unless B-cell recovery is proven.
* 12. Received immunosuppressants and other small molecule drugs within 3 days before infusion.
* 13. Use of any other clinical research drugs within 4 weeks before infusion. However, if the study treatment is ineffective or the disease progresses during the study period, and at least 3 half-lives have elapsed before screening, enrollment is allowed.
* 14. The patient has received live vaccines or live therapeutic infectious pathogens within 2 weeks before infusion.
* 15. The presence of chronic and active hepatitis B (excluding HBV-DNA levels below 500IU/ml), hepatitis C (HCV), human immunodeficiency virus (HIV) infection, or syphilis infection;
* 16. Active infection exists, requiring intravenous antibiotic therapy or hospitalization;
* 17. Patients who have undergone major surgery other than diagnosis or biopsy within 4 weeks before infusion, or are expected to undergo major surgery during the study period; note: patients who plan to undergo surgical procedures under local anesthesia can participate in the study.

Kyphoplasty or vertebroplasty are not considered major surgery;

* 18. Obvious evidence of cardiovascular disease as follows: a. N-terminal pro-B-type natriuretic peptide (NT-proBNP) > 8500ng/L; b. New York Heart Association (NYHA) classification of heart failure as III or IV; c. Patients who have received inpatient treatment for unstable angina or myocardial infarction within 6 months before the first dose, or who have received percutaneous coronary intervention and have received the latest stent placement within 6 months, or who have received coronary artery bypass grafting within 6 months;
* 19. Individuals who have known allergies, hypersensitivity reactions, intolerances, or contraindications to any component of V001-BCMA, or who have previously experienced severe allergic reactions.
* 20. Those who were deemed unsuitable for infusion or otherwise unsuitable for participation in the study by the researchers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events of V001-BCMA single infusion. | At Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For all participants

SECONDARY OUTCOMES:
BILAG-2004 Scale Score | At baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  The BILAG-2004 index assesses disease activity in systemic lupus erythematosus (SLE) to guide treatment. It evaluates nine organ systems separately, grading each from A to E based on clinical features: A (severe, requiring aggressive therapy), B (moderate), C (mild), D (previous involvement), and E (no involvement). Its focus is on tracking changes per system for targeted management.
PGA | At baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  Physician Global Assessment. PGA score is used to assess the disease activity status of patient by physician. PGA min-max(0-3, the higher score represents the worse result)
SF-36 | At baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  The 36-Item Short Form Health Survey. For SLE and AAV. SF-36 score min-max(0-100,the higher score represents the better result)
DORIS score | At Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  The DORIS score defines remission criteria in systemic lupus erythematosus (SLE), guiding treatment goals and trial endpoints. Its core assessment includes: 1) clinical SLEDAI=0; 2) Physician Global Assessment (PGA)<0.5; 3) prednisone ≤5mg/day; 4) stable immunosuppressive/biologic therapy. It also requires stable/improved serology and sustained duration of remission.
LLDAS | At Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  The LLDAS defines a "low disease activity state" in SLE, a key treatment target linked to better long-term outcomes. Core criteria include: 1) SLEDAI-2K ≤4; 2) no new disease activity; 3) Physician Global Assessment (PGA) ≤1.0; 4) prednisone ≤7.5mg/day; 5) stable immunosuppressive/biologic doses.
Renal function response | At Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  Only for LN patients
Cmax | Baseline, Day 2, Day 6, Day 10, Day 14, Day 21, Day 28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24
  For all subjects. Parameters of CAR copy number
Tmax | Baseline, Day 2, Day 6, Day 10, Day 14, Day 21, Day 28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24
  For all subjects
AUC0-28d | Baseline, Day 2, Day 6, Day 10, Day 14, Day 21, Day 28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24
  For all subjects
AUC0-90d | Baseline, Day 2, Day 6, Day 10, Day 14, Day 21, Day 28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24
  For all subjects
Tlast | Baseline, Day 2, Day 6, Day 10, Day 14, Day 21, Day 28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24
  For all subjects
24-hour urine protein | Baseline, Day 2, Day 6, Day 10, Day 14, Day 21, Day 28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24
  Only for LN
UPCR | Baseline, Day 2, Day 6, Day 10, Day 14, Day 21, Day 28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24
  UPCR (Urine Protein-to-Creatinine Ratio) is a key index to measure assessing treatment response in lupus nephritis.
Proportion of CAR-T cells in T cells | baseline、Day 2、Day 6、Day 10、Day 14、Day 21、Day 28 after infusion
  For all subjects
serum sBCMA level | Screening period, baseline, Day 14, Day 28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 post-infusion.
  BCMA expression levels of memory B cells and plasma blast cells in peripheral blood
Time to disease recurrence | through study completion (at most 52 weeks)
  For IgG4-RD. Defined as the number of days between the day of infusion and the date of first treatment for IgG4-RD recurrence, as determined by a clinical professional, during the follow-up period
Changes in lymphocyte subpopulations | Screening period, Day 14, Day 28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion, and at recurrence
  For all subjects
Proportion of patients with improved disease activity (IgG4-RD RI) | Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For IgG4-RD. Improvement is defined as a decrease of ≥2 from the baseline disease activity score
annualized recurrence rate | through study completion, an average of 1 year
  For IgG4-RD
The proportion of subjects who achieved complete remission without relapse at week 52 | at week 52
  For IgG4-RD
Change in CRISS-25 score from baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For systemic sclerosis. The score of CRISS-25 min-max(0-1.0, the higher score represents the better result)
Change in forced vital capacity (FVC) (mL) from baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For systemic sclerosis
Change in mRSS from baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For systemic sclerosis. The score of mRSS min-max(0-51, the higher score represents the worse result)
Change from baseline in Quantitative Interstitial Lung Disease (QILD) imaging score | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For systemic sclerosis. The min-max score (0-100%, the higher score represents the worse result)
Change from baseline in Quantitative Lung Fibrosis (QLF) imaging score | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For systemic sclerosis. The min-max score (0-100%, the higher score represents the worse result)
Changes in Scleroderma Patient Skin Report (SSPRO) compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For systemic sclerosis.The min-max score (0-108, the higher score represents the worse result)
Changes in Scleroderma Clinical Trial Consortium Damage Index (SCTC-DI) compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For systemic sclerosis. The min-max score (0-55, the higher score represents the worse result)
Changes in EUSTAR activity index scores compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For systemic sclerosis The min-max score (0-10, the higher score represents the worse result)
Changes in Capillaroscopic skin ulcer risk index (CSURI) compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For systemic sclerosis. CSURI is a continuous variable; the higher the score, the greater the ulcer risk.
Changes in Gastrointestinal questionnaire scores of the University of California, Los Angeles Scleroderma Clinical Trial Alliance compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For systemic sclerosis.The min-max score (0-3, the higher score represents the worse result)
Changes in serum SSc-related antibodies compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For systemic sclerosis
Changes in Muscle Strength Score (MRC) compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For idiopathic inflammatory myopathies. The min-max score (0-60, the higher score represents the better result)
The changes in total improvement score (TIS) compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For idiopathic inflammatory myopathies. The min-max score (0-100, the higher score represents the better result)
Changes in lesion size and severity index (CDASI) compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For idiopathic inflammatory myopathies. The CDASI is a core instrument for assessing the severity of cutaneous dermatomyositis. It consists of two independent subscales: Activity (scored 0-100, with higher scores indicating worse status) and Damage (scored 0-32, with higher scores indicating worse status).
Physician's overall disease activity score | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For idiopathic inflammatory myopathies. The min-max score (0-10, the higher score represents the worse result)
Changes in Manual Muscle Testing 8 (MMT8) compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For idiopathic inflammatory myopathies. The min-max score (0-150, the higher score represents the better result)
Changes in Expanded Myositis Disease Activity Index (EMDA) compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For idiopathic inflammatory myopathies. The min-max score (0-10, the higher score represents the worse result)
Changes in MDAAT score compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For idiopathic inflammatory myopathies. the overall score of extramuscular disease activity was assessed using the MDAAT scoring tool. The min-max score (0-60, the higher score represents the worse result)
Myositis Core Set Measures | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For idiopathic inflammatory myopathies
the remission rate of myositis (defined as an increase in TIS of ≥20, ≥40, and ≥60 points) was assessed according to the 2016 ACR/EULAR criteria for myositis remission | Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For idiopathic inflammatory myopathies
Time to improvement (TIS≥20, ≥40 and ≥60) | up to 52 weeks
  For idiopathic inflammatory myopathies
Duration of remission (time from clinical remission to deterioration/time from remission to first recurrence) | up to 52 weeks
  For idiopathic inflammatory myopathies
Changes in myositis specific antibodies and myositis associated antibodies in serum compared to baseline after injection | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For idiopathic inflammatory myopathies
Changes in ILD on CT imaging compared to baseline (only for patients with ILD at baseline) | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For idiopathic inflammatory myopathy patients with ILD in the baseline period
Pulmonary function examination evaluates changes in ventilation and diffusion function compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For idiopathic inflammatory myopathies. Pulmonary function examination can comprehensively evaluate the ventilation function, air exchange function, and airway responsiveness of the lungs, which is of great significance for the diagnosis, condition evaluation, and efficacy judgment of respiratory diseases
Myositis specific antibody levels | Screening period, baseline, Day 14, Day 28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 post-infusion.
  For idiopathic inflammatory myopathies
Myositis related antibody levels | Screening period, baseline, Day 14, Day 28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 post-infusion.
  For idiopathic inflammatory myopathies
The proportion of subjects who maintained remission | Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For AAV
duration of response | Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For AAV
Changes in Vasculitis Damage Index (VDI) scores compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For AAV
Changes in quality of life (SF-36 V2 scale) scores compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For AAV. The min-max score (0-100, the higher score represents the better result)
Changes in Disease Scope Index (DEI) compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For AAV. The min-max score (0-21, the higher score represents the worse result)
Changes in Five Factor Score (FFS) compared to baseline | At Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 after infusion
  For AAV. The min-max score (0-5, the higher score represents the worse result)

OTHER OUTCOMES:
Virus Leak Detection | baseline、Day2、Day4、Day6、Day8、Day10、Day14、Day21、Day28
  For all subjects. Collect blood, saliva, urine, and fecal samples for cryogenic storage and detect any potential leaks. Collect blood, saliva, urine, and fecal samples to detect virus levels and determine if there is a carrier virus leak
immunogenicity | baseline、Day28、Month3，Month6，Month9，Month12，Month18，Month24 post infusion
  For all subjects. Detecting anti CAR antibodies in patient serum using bridging ELISA or flow cytometry
Single-cell sequencing | During the screening period, at either 3 months or 6 months, the specific timing of the test will be determined by the researcher
  For all subjects. Collect peripheral blood from patients and perform single-cell sequencing. Droplet platforms (such as 10 × Genomics) are the most commonly used scRNA seq platforms. The platform places single cells into water in oil droplets containing gel beads through the microfluidic chamber. gel beads have mRNA capture primers, unique molecular barcodes, and enzyme/reagent mixtures required for cell lysis and reverse transcription. After reverse transcription of transcription information to obtain cDNA, high-throughput sequencing can be performed through PCR amplification and library preparation.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China